CLINICAL TRIAL: NCT00338572
Title: Sympathetic Nervous System Regulation of Cell Adhesion
Brief Title: Effect of Exercise and Diet on Inflammation in Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul J. Mills, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 380; R01HL057265 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Inflammation; Blood Pressure, High
MeSH Terms: conditions — Hypertension; Inflammation | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 12-week exercise program
  Interventions: Behavioral: Exercise Program
- 2 (Experimental): 12-week combined exercise and diet program
  Interventions: Behavioral: Combined Exercise and Diet Program
- 3 (No Intervention): Non-intervention group

INTERVENTIONS:
Behavioral: Exercise Program — Participants in the exercise group will receive a 12-week membership to the YMCA and will meet with a personal trainer twice a week. They will be encouraged to exercise on their own for an additional 3 to 4 days per week. Participants will also be provided with a pedometer, which will track the number of steps they take each day.
  Arms: 1
Behavioral: Combined Exercise and Diet Program — Participants in this group will receive a 12-week membership to the YMCA and will meet with a personal trainer twice a week. They will be encouraged to exercise on their own for an additional 3 to 4 days per week. Participants will also be provided with a pedometer, which will track the number of steps they take each day. They will meet with a dietician and will be encouraged to reduce their caloric intake by incorporating low-fat, high-fiber foods into their diet.
  Arms: 2

SUMMARY:
In addition to high blood pressure, hypertension is characterized by inflammation, which is the body's response to injury or infection. Inflammation has been found to cause plaque formation on artery walls. This study will compare the effect of an exercise program versus a combined exercise and diet program on reducing inflammation in hypertensive individuals.

DETAILED DESCRIPTION:
Hypertension is characterized by high blood pressure, as well as by inflammation and increased adhesion among blood cells. Inflammation may play an important role in atherosclerosis, which involves the build up of fatty deposits on the inside wall of arteries. Pharmacological treatment for hypertension successfully reduces blood pressure. However, it has limited effectiveness for reducing the associated inflammation. Losing weight and increasing physical activity have been shown to reduce general inflammation, but more research is needed to determine their effect on inflammation that is directly related to hypertension. The purpose of this study is to evaluate the effectiveness of an exercise program versus a combined exercise and diet program at reducing inflammation and cell adhesion in hypertensive individuals.

This study will enroll inactive and overweight hypertensive individuals. Participants will be randomly assigned to a 12-week exercise program, a 12-week combined exercise and diet program, or a non-intervention group. At study entry, participants will take part in a speech stressor task, a VO2 peak exercise test, and an exercise treadmill test. During the speech stressor task, participants will be videotaped while they talk about potentially stressful situations. Prior to and following the speech task, blood will be collected, blood pressure and heart rate will be recorded, and standardized questionnaires will be completed to assess anger, anxiety, and stress levels. The two exercise tests will occur within 5 days of each other and both will involve running on a treadmill. Heart rate, respiratory rate, and physical activity intensity will be monitored; heart activity will be measured by an electrocardiogram (ECG). Blood will be collected at various times during the testing procedures to measure levels of inflammation biomarkers, including C-reactive protein (CRP) and white blood cells. Perceived exertion and stress levels will also be assessed.

Participants in the exercise intervention will receive a 12-week membership to the YMCA and will meet with a personal trainer twice a week. They will be encouraged to exercise on their own for an additional 3 to 4 days per week. Participants will also be provided with a pedometer, which will track the number of steps they take each day. Participants in the diet program will meet with a dietician and will be encouraged to reduce their caloric intake by incorporating low-fat, high-fiber foods into their diet. Throughout the study, participants will have regular follow-up phone calls with study staff and meetings with their personal trainer and/or dietician to ensure that they are adhering to their assigned program. At the end of 12 weeks, participants will return for a repeat speech stressor task, a VO2 peak exercise test, and an exercise treadmill test. Participants in the non-intervention group will then be assigned to either the exercise program or combined exercise and diet program.

ELIGIBILITY:
Inclusion Criteria:

* Unmedicated hypertension with blood pressure greater than 140/90 mm Hg but less than 175/104 mm Hg
* Body mass index (BMI) of 23.5 to 34
* Relatively inactive, as defined by the Leisure Time Exercise Questionnaire
* Willing and able to participate in the assigned study group
* Postmenopausal women not on hormone replacement therapy (HRT) and premenopausal women

Exclusion Criteria:

* Abnormal echocardiogram
* Recent stroke or significant brain impairment
* Current psychiatric disease
* History of psychosis or major depression
* Currently taking psychotropic drugs
* Currently taking any medications (e.g., anti-inflammatory medications) other than antihypertensives (which will be tapered)
* Current drug and/or alcohol abuse
* Consumes more than 600 mg of caffeine per day
* Diabetes
* Congestive heart failure
* Bronchospastic pulmonary disease
* History of heart attacks
* Known secondary high blood pressure
* Angina
* History of life-threatening arrhythmias
* History of kidney damage
* Current participation in regular or structured exercise classes, or regular physical exercise in the 6 months prior to study entry
* Inability to perform moderate to vigorous intensity exercise
* Current participation in a diet
* High blood pressure, only when measured in a doctor's office (i.e., "white coat hypertension")
* Arthritis, exertional asthma, or any other disorder likely to be made worse by exercise
* Pregnant

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2006-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
CRP | Measured at 4 years
Interleukin-6 (IL-6) | Measured at 4 years
Tumor necrosis factor-alpha (TNF-alpha) | Measured at 4 years
Soluble intercellular adhesion molecule-1 (sICAM-1) | Measured at 4 years
SE-selectin | Measured at 4 years
Leukocyte CD11a expression | Measured at 4 years
Leukocyte CD11b expression | Measured at 4 years
Leukocyte activation | Measured at 4 years
Peripheral blood mononuclear cell chemotaxis | Measured at 4 years

SECONDARY OUTCOMES:
Physical fitness | Measured at 4 years
Weight | Measured at 4 years
Blood pressure | Measured at 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Mills, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States